CLINICAL TRIAL: NCT05334875
Title: Repeatability of Electroretinogram and Visual Evoked Potential in Clinical Practice
Brief Title: Repeatability of Electroretinogram and Visual Evoked Potential
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelshafy, Lecturer of Ophthalmology, Benha University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RC 8-22
Record Dates: First submitted 2022-04-07; First posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Retinal Disease; Visual Impairment; Vision Disorders
Keywords: Electroretinogram; Visual evoked potential
MeSH Terms: conditions — Retinal Diseases; Vision Disorders | interventions — Electroretinography; Evoked Potentials, Visual

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electroretinogram test (ERG) (Active Comparator): ERG test will be done for each subject twice and compare the results to assess repeatability of the test.
  Interventions: Diagnostic Test: Electroretinogram (ERG)
- Visual evoked potential test (VEP) (Active Comparator): VEP test will be done for each subject twice and compare the results to assess repeatability of the test.
  Interventions: Diagnostic Test: Visual evoked potential (VEP)

INTERVENTIONS:
Diagnostic Test: Electroretinogram (ERG) — Applying electrodes to assess retinal function
  Arms: Electroretinogram test (ERG)
Diagnostic Test: Visual evoked potential (VEP) — Applying electrodes to assess visual pathway function
  Arms: Visual evoked potential test (VEP)

SUMMARY:
To assess repeatability of electroretinogram and visual evoked potential in clinical practice

DETAILED DESCRIPTION:
To assess repeatability of electroretinogram in evaluation of retinal function and visual evoked potential in evaluation of visual pathway in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Normal subjects visit banha university hospital seeking regular checkup and subjects asked for ERG and VEP as a pre-occupational examination.

Exclusion Criteria:

* Patients previously diagnosed with any retinal disease or visual pathway disease that may affect ERG and VEP tests.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Repeatability of ERG amplitude. | Changes from baseline measurements and at one week.
  ERG amplitude measured in nano volt (nV).

SECONDARY OUTCOMES:
Repeatability of ERG latency. | Changes from baseline measurements and at one week.
  Latency of ERG measured by millisecond (msec).

OTHER OUTCOMES:
Repeatability of VEP amplitude. | Changes from baseline measurements and at one week.
  VEP amplitude measured in nano volt (nV).
Repeatability of VEP latency. | Changes from baseline measurements and at one week.
  Latency of VEP measured by millisecond (msec).

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A Abdelshafy, MD, Study Chair — Benha University
Locations (1):
- Ahmed Abdelshafy Tabl, Banhā, Benha, Egypt